CLINICAL TRIAL: NCT04458727
Title: Auswertung Von Multi-modalen unterstützenden Maßnahmen in Der Ambulant Kardiologischen Rehabilitation Bei Patienten Mit Einer kardiovaskulären Erkrankung
Brief Title: Evaluation of Multi-modal Supportive Actions in Outpatient Cardiac Rehabilitation in Subjects With Cardiovascular Disease
Acronym: EPICURE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: AIT Austrian Institute of Technology GmbH (Other)
Collaborators: Cardiomed Kardiologisches Rehabilitationszentrum GmbH Linz (Unknown); PKA Private Krankenanstalt Wels Betriebs Gesellschaft mit b. H. (Unknown); Gemeinnützige Salzburger Landeskliniken Betriebsgesellschaften (Unknown); Medreha GmbH (Unknown); ZARG - Zentrum für ambulante Rehabilitation Graz GmbH (Unknown); REHAmed-tirol GmbH Innsbruck (Unknown); Universität Innsbruck (Unknown)
Responsible Party: Sponsor
Other Study IDs: EPICURE
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Evaluation of Multi-modal Supportive Actions in Outpatient Cardiac Rehabilitation in Subjects With Cardiovascular Disease
Keywords: rehabilitation; cardiovascular disease; outpatient cardiac rehabilitation
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients who used supportive measures during home training
- patients who did not use supp. measures during home training

SUMMARY:
Cariovascular diseases (CVD) are the most common cause of death worldwide with high micro- as well as macro-economic burden. Several modifiable risk factors increase the probability of contracting a CVE. These risk factors can be positively influenced by a cardiac rehabilitation measure (CR), which has been shown to reduce mortality in CVD patients and to reduce the economic burden. An increase in physical activity and performance are central goals in CR, as they have a positive effect on several cardiovascular risk factors and correlate strongly with a reduction in mortality in CVD patients. These goals can be achieved in most CVD patients but can only be achieved by a modification of lifestyle.

In order to positively influence this lifestyle modification beyond the duration of the CR measure and thus in the long term, CR Phase II should begin as soon as the patient fulfils one of the well-defined inclusion criteria. CR Phase II can be carried out as an inpatient or outpatient procedure and depends on the patient's state of health, personal preference and availability of an outpatient CR facility in the vicinity of the patient. In the Austrian healthcare system, inpatient CR and thus differs from other European countries. After completion of phase II, the patient is offered an outpatient phase III with weekly visits to the outpatient CR facility, so that lifestyle changes achieved at short notice can be sustainably maintained.

For the secondary prevention of the CVD beyond the CR measure recommend international guidelines a physical activity of ≥ 150 min with moderate intensity or ≥ 60 to 75 min high intensity per week. The current study situation allows the statement that a greater benefit can be expected from more physical activity and that the training should be personalized and highly titrated. Patients in advanced stages of CVD and very inactive patients, defined as <14 mets h/week, achieve the greatest health benefit from increased physical activity. Despite the well-studied benefits, even adherence to the above minimum recommendations for CVD patients after completion of CR is low. This deficit has been addressed in the latest European prevention guideline and recommended that patients i) set clearly defined goals, ii) exercise in the iii) Identify obstacles on the way to achieving the goals so that lifestyle changes are effective and sustainable and the benefits of physical activity can be achieved and maintained.

The planned study will investigate the effect of multi-modal support measures to help patients during the home training phase and their influence on the patients' lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Participation rehabilitation phase III new
* Documented cardiovascular disease
* Signed informed-consent

Exclusion Criteria:

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who undergo the final examination for OUT-III at one of the outpatient rehabilitation facilities participating in the study are checked by the examining physician for the above-mentioned inclusion and exclusion criteria. Patients will be included if they are willing to participate and sign the consent form.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2020-09-09 (Estimated); Study Completion 2020-09-09 (Estimated)

PRIMARY OUTCOMES:
The change of maximal workload during ergometry pre and post home-training | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiomed Kardiologisches Rehabilitationszentrum GmbH Linz, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: Undecided